CLINICAL TRIAL: NCT04678804
Title: Connective Tissue Graft Versus Collagen Matrix. A 3D Digital Soft Tissue Thickening Analysis in Mucogingival Surgery: a 6 Months Follow-up Pilot Study
Brief Title: Connective Tissue Graft Versus Collagen Matrix.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Prof Elena Calciolari, Researcher, University of Parma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 808/2019/DISP/UNIPR
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Gingival Diseases
MeSH Terms: conditions — Gingival Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Matrix Graft Group (Experimental): patients treated with Porcine Derived Volume Stable Matrix
  Interventions: Procedure: Mucogingival surgery for single recession coverage
- Autogenous ctg group (Other): patients treated with autologous tissue
  Interventions: Procedure: Mucogingival surgery for single recession coverage

INTERVENTIONS:
Procedure: Mucogingival surgery for single recession coverage — The control group will be treated with a coronally advanced flap with vertical incisions (CAF) associated to an autologous connective tissue graft. The graft will be harvested from the palate in the area apical to the gingival margin of the second molar with an epithelial-connective harvesting technique to obtain a connective graft of 1 mm in thickness.
  Subsequently, the graft will be shaped in order to match height and width of the recipient site on the recession according to the technique proposed by Zucchelli in 2003. The test group will receive the same flap design with the same technique, then the porcine derived xenogeneic graft will be shaped in order to match height and width of the recipient site on the recession. In particular, the matrix will be reduced in thickness as suggested by the manufacturer to obtain a standardized thickness of 3 mm.

SUMMARY:
Despite the potential role of soft tissue thickness in maintaining gingival margin stability, the existing literature has mainly focused on investigating the effect of different surgical techniques on recession coverage percentage, without taking into account the changes in tissue thickness and biotype in the surgical area. Hence, this study aims to compare threedimensional scans of gingival recessions treated either with CAF+CTG or with CAF+PDCM by the use of a dedicated superimposition software at different healing timepoints.

The primary outcome is to assess the change in mm3 and the distribution pattern of soft tissue thickening in the surgical area between autologous and heterologous grafts at 1, 3, and 6 months post-surgery. The secondary outcomes are: the complete root coverage at 6 months post surgery and Patients' Reported Outcomes (PROMS) measured with oral impact on daily performances (OIDP questionnaire) and on the evaluation of patients' perception about therapy.

DETAILED DESCRIPTION:
This is a pilot study and will include 8 visits over a minimum period of 25 weeks. The trial will follow the recommendations of the Consolidated Standards of Reporting Trials (CONSORT) statement and will be registered in clinicaltrials.gov after the obtainment of the relevant approval from ethics committee. All the relevant authorization (Ethical committee, Insurance) will be obtained before study initiation. Study population: 12 patients will be recruited in the new patient and follow-up clinics which run every week at the Centre of Dentistry of University of Parma.

Main inclusion criteria:

* Systemically healthy males and females ≥ 18 years old
* Willingness to read and sign a copy of the Informed Consent Form after reading the Patient Information Sheet, and after the nature of the study has been fully explained
* Clinical evidence of a single gingival recession (RT1, RT2)
* Full mouth bleeding and plaque scores (FMBS and FMPS) < 20% recorded
* Non-surgical treatment completed within 6 months prior to assessment for eligibility

Main inclusion criteria:

* Medical history that includes diabetes or hepatic or renal disease, or other serious medical conditions or transmittable diseases (e.g. cardiovascular disease or AIDS).
* Antibiotic, anti-inflammatory or anticoagulant therapy during the month preceding the baseline exam.
* History of alcohol or drug abuse.
* Smoking ≥10 cigarettes a day
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results).
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial.
* Taking medications that might induce gingival overgrowth (e.g. calcium antagonists)

Study visits:

Visit 1 - Baseline -

* Informed consent, medical/dental history and demographics
* Record concomitant medications and smoking history
* Periodontal assessment by a blind and calibrated examiner, consisting of full mouth PPD, REC, BOP, mobility and furcation involvement will be recorded. PPD, REC, plaque and BOP will be recorded at 6 sites per tooth.
* Intra-oral 3D scan in the area selected for the study
* PROMs assessment (OIDP and Global changes in Quality of Life)
* Pre-treatment hygiene phase, including supragingival scale and polish of all teeth and oral hygiene instructions
* Randomization to one of the two treatment groups by the study co-ordinator. The treatment allocation will be concealed in an opaque envelope. A treatment visit will be scheduled within the following 6 weeks.
* Standardized high definition intraoral photos Visit 2 - Surgical intervention - (within 12 weeks from Visit 1)
* Query to update medical/dental history and record adverse events and/or concomitant medications
* Study treatment according to randomization (CTG or PDCM)
* Post-surgical instructions
* Standardized high definition intraoral photos Visit 3 - 7 days follow up - (within 7d + 2d from Visit 2)
* Standardized high definition intraoral photos
* Visual assessment of gingival healing
* PROMs assessment Visit 4 - 14 days follow up - (within 14d ± 3d from Visit 2)
* Standardized high definition intraoral photos
* Visual assessment of gingival healing
* PROMs assessment
* Sutures removal Visit 5 - 21 days follow up - (within 21d ± 3d from Visit 2)
* Standardized high definition intraoral photos
* Visual assessment of gingival healing
* PROMs assessment Visit 6 - 30 days follow up - (within 30 ± 3d from Visit 2)
* Standardized high definition intraoral photos
* Visual assessment of gingival healing
* PROMs assessment
* Intraoral 3D scan Visit 7 - 3 months follow up - (within 3 months ± 1w from Visit 2)
* Standardized high definition intraoral photos
* Visual assessment of gingival healing
* Intraoral 3D scan Visit 8 - 6 months follow up - (within 6 months ± 1w from Visit 2)
* Standardized high definition intraoral photos
* Visual assessment of gingival healing and complete root coverage (UNC-15 probe)
* Intraoral 3D scan Study randomization and treatment allocation: A specifically designed locked computer software program will be used to randomly assign patients to one of two study groups: the control group of 6 patients treated with CAF+CTG and the test group of 6 patients treated with CAF+PDCM (Fibrogide). The allocation result will be kept in a locked computer file that will not not accessible to examiners and practitioners. The operator will be informed about the patient's allocation on the day of the intervention. Surgical procedures: The control group will be treated with a bilaminar technique where a coronally advanced flap with vertical incisions (CAF) according to the technique described by Langer in 1885 is associated to an autologous connective tissue graft. The graft will be harvested from the palate in the area apical to the gingival margin of the second molar with an epithelial-connective harvesting technique to obtain a connective graft of 1 mm in thickness.

Subsequently, the graft will be shaped in order to match height and width of the recipient site on the recession according to the technique proposed by Zucchelli in 2003. The test group will receive the same flap design with the same technique, then the porcine derived xenogeneic graft will be shaped in order to match height and width of the recipient site on the recession. In particular, the matrix will be reduced in thickness as suggested by the manufacturer to obtain a standardized thickness of 3 mm. Patients will be instructed to avoid any mechanical trauma or tooth brushing in the surgical sites for 3 weeks. They will be instructed to take painkiller medications if necessary.

Chlorhexidine 1% gel applications will be prescribed three times per day for 2 weeks. Sutures will be removed after 14 days. Three weeks after surgery, patients will be instructed to resume gently mechanical tooth cleaning with an extra-soft toothbrush. 3D imaging: Digital impressions obtained with an intraoral scanner (Carestream CS 3600, Carestream Dental, Atlanta GA, USA) will be employed to evaluate soft tissue volumetric changes before treatment (T0), at 1 month (T1) and at 3 months (T2) and 6 months (T3) after surgery. The 6 months follow-up visit was chosen as the endpoint of this study in consideration of the complete resorption time of the PDCM as described by the manufacturer.

Digital 3D images will be converted info STL files. STL is a file format created to describe only the surface geometry of a three-dimensional object without any representation of color, texture or other common CAD model attributes. A dedicated software (MeshLab, ISTI-CNR, Rome, Italy) with a professional digital environment that allows the operator to import, open and manage STL files will then be employed to analyze the three STL files obtained at different timepoints (T0, T1, T2, T3) by a blind operator. More specifically, the software will accurately superimpose the scans by using a minimum of 4 reference points identified by a collimation process. Then the area of interest (an area of 10 x 10 mm, apical to the CEJ) will be isolated and the difference in volume (mm3) will be calculated by the software. In addition, the software will also return an analysis of the thickening distribution pattern in the area of interest. It is important to emphasise that this protocol for 3D image analysis has been already validated and succesfully tested in ten pilot cases. (FIG 1,2,3,4) PROMs: The OIDP is a well validated and frequently used PROM in studies of oral health. It is a composite measure of the impacts of oral health on the quality of life of people (eating, speaking, cleaning teeth, going out, relaxing, smiling, major work or role, emotional stability, social contact). The overall OIDP score ranges from 0 to 100, with higher scores indicating worse quality of life. Furthermore, when an oral impact is reported, the patient is further asked which oral condition was responsible for that impact. In the 7, 14 and 30 days follow-up visits, we will also evaluate patient perception about therapy. More specifically, the extent of discomfort and/or pain experienced will be evaluated using a 100-mm horizontal visual analog scale (VAS). The anchors for each end of the scales will be designated as none and extreme. Patients will be also instructed to quantify the analgesic medication taken. In addition, the extent of discomfort, root hypersensitivity, oedema, hematoma, high fever, and interference in daily activities during the first posttherapy week will be evaluated in the same way. Root coverage assessment: The complete root coverage measured as the residual distance from the gingival margin to the CEJ will be recorded with a UNC-15 periodontal probe by a calibrated blind examiner at the 6 months follow-up appointment. Sample size calculation: Since this can be considered as a pilot study (no other studies in the literature have used this 3D approach to evaluate changes in tissue thickness), the sample size calculation was based on previous studies' results in this field and on the investigators' experience. We speculated that 10 patients per group would allow to collect enough data to power future trials (if needed). A 20% drop-out rate was also considered, thus leading to a total of twelve patients (6 per group) to be enrolled for the study. Outcomes and Statistics: The primary outcome of the study is to analyze and measure the soft tissue thickness modifications in the area of the graft with the three-dimensional superimposition technique. The measurement will be performed in cubic millimeters and the distribution will be analyzed with a colorimetric graphic map. The modifications will be compared between groups and between timepoints with an inter/intra group analysis.

The secondary outcomes consider linear measurements and PROMs. In addiction, the superimposition software will be used to assess the thickness increase at six months. More specifically, two-dimensional linear measurements will be performed perpendicular to the alveolar crest along the vertical axis of the tooth from the center of the gingival and will be repeated each mm for 10 mm in apical direction (Gonzales-martin 2014). The modifications will be compared between groups and between timepoints with an inter/intra group analysis.

Patients' Reported Outcomes (PROMS) will be measured with oral impact on daily performances (OIDP questionnaire) and on the evaluation of patients' perception about therapy. Clinical measurements will be performed by a blind calibrated operator.

T-Test and Factorial Effect Anova Test will be performed in order to statistically analyze the results in the test and control groups at different timepoints.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy males and females ≥ 18 years old

* Willingness to read and sign a copy of the Informed Consent Form after reading the Patient Information Sheet, and after the nature of the study has been fully explained
* Clinical evidence of a single gingival recession (RT1, RT2)
* Full mouth bleeding and plaque scores (FMBS and FMPS) < 20% recorded
* Non-surgical treatment completed within 6 months prior to assessment for eligibility

Exclusion Criteria:

* Medical history that includes diabetes or hepatic or renal disease, or other serious medical conditions or transmittable diseases (e.g. cardiovascular disease or AIDS).

  * Antibiotic, anti-inflammatory or anticoagulant therapy during the month preceding the baseline exam.
  * History of alcohol or drug abuse.
  * Smoking ≥10 cigarettes a day
  * Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results).
  * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial.
  * Taking medications that might induce gingival overgrowth (e.g. calcium antagonists)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Soft tissue modifications | 6 months
  to analyze and measure the soft tissue thickness modifications in the area of the graft with the three-dimensional superimposition technique. The measurement will be performed in cubic millimeters and the distribution will be analyzed with a colorimetric graphic map. The modifications will be compared between groups and between timepoints with an inter/intra group analysis.

SECONDARY OUTCOMES:
PROMS | 6 months
  Patients' Reported Outcomes (PROMS) will be measured with oral impact on daily performances (OIDP questionnaire) and on the evaluation of patients' perception about therapy. Clinical measurements will be performed by a blind calibrated operator.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Calciolari, DDS, Principal Investigator — Researcher
Locations (1):
- Centro Universitario di Odontoiatria, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cairo F, Nieri M, Cincinelli S, Mervelt J, Pagliaro U. The interproximal clinical attachment level to classify gingival recessions and predict root coverage outcomes: an explorative and reliability study. J Clin Periodontol. 2011 Jul;38(7):661-6. doi: 10.1111/j.1600-051X.2011.01732.x. Epub 2011 Apr 20. PMID 21507033
- [Result] Thoma DS, Zeltner M, Hilbe M, Hammerle CH, Husler J, Jung RE. Randomized controlled clinical study evaluating effectiveness and safety of a volume-stable collagen matrix compared to autogenous connective tissue grafts for soft tissue augmentation at implant sites. J Clin Periodontol. 2016 Oct;43(10):874-85. doi: 10.1111/jcpe.12588. Epub 2016 Aug 12. PMID 27310522
- [Result] Langer B, Langer L. Subepithelial connective tissue graft technique for root coverage. J Periodontol. 1985 Dec;56(12):715-20. doi: 10.1902/jop.1985.56.12.715. PMID 3866056
- [Result] Zucchelli G, Amore C, Sforza NM, Montebugnoli L, De Sanctis M. Bilaminar techniques for the treatment of recession-type defects. A comparative clinical study. J Clin Periodontol. 2003 Oct;30(10):862-70. doi: 10.1034/j.1600-051x.2003.00397.x. PMID 14710766